CLINICAL TRIAL: NCT05898100
Title: Effects of The Virtual Reality "Dream" Game on Anxiety During Dental Procedures in Children (VR-TOOTH): A Pilot Randomized, Controlled Trial
Brief Title: Virtual Reality Distraction for Dental Anxiety (PILOT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Sylvie Le May, Principal Investigator, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VR-TOOTH-PILOT
Record Dates: First submitted 2023-04-04; First posted 2023-06-12 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Dental Anxiety; Dental Phobia; Dental Trauma; Dental Diseases
MeSH Terms: conditions — Stomatognathic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Reality Distraction (Experimental): Use of virtual reality (VR) during dental procedure.
  Interventions: Device: Virtual Reality Distraction
- Standard Treatment (Active Comparator): Dental Clinic's standard treatment during dental procedure.
  Interventions: Behavioral: Dental Clinic's Standard Treatment

INTERVENTIONS:
Device: Virtual Reality Distraction — The experimental group will receive the VR video game Dream designed specifically for this study. Pharmaceutical treatment during the procedure such as the use of injected local anesthesia will be used if the procedure requires. Children will be able to play for the entire duration of the dental procedure. Dream aims at reducing anxiety in children aged 6 to 17 years old by mean of immersive distraction. The VR headset offers children with the ability of viewing the game they are playing in real time while simultaneously obstructing the partial view they would normally have of the procedure. In the event of non-cooperation during the appointment, any re-take or re-scheduling appointments will be compiled by the resident dentist. One parent will be allowed in the room during the dental procedure and their presence will be recorded.
  Arms: Virtual Reality Distraction
Behavioral: Dental Clinic's Standard Treatment — The control group will only receive a care-as-usual approach. This includes a television mounted on the wall showing cartoons and the use of pharmaceutical treatment during the procedure such as the use of injected local anesthesia. In the event of non-cooperation during the appointment, any re-take or re-scheduling appointments will be compiled by the resident dentist. One parent will be permitted to be present in the room during the procedure as part of the clinic's usual protocol and their presence will be recorded. Children allocated to the control group will be offered the possibility to try the VR game after the study period if they choose so.
  Arms: Standard Treatment

SUMMARY:
Introduction. Dental fear and anxiety (DFA) is a condition that affects approximately a quarter of children and adolescents. Lack of patient cooperation due to DFA can create an environment of stress, often obligating dentists to end appointments prematurely. Virtual reality use could improve DFA in children with special health care needs (SHCN) undergoing dental procedures.

Aim. Assess the feasibility and acceptability of VR immersion as a tool to reduce dental fear and anxiety in pediatric special needs patients undergoing dental procedures and gain insight on parents and healthcare providers perspectives on the use of VR during dental appointments.

Methods. This pilot randomized controlled trial study will follow a parallel design including two groups: A control group (clinic's standard care) and an experimental group (virtual reality). Twenty participants will be randomized to either group. Recruitment will be carried out at the dental clinic of the Centre Hospitalier Universitaire Sainte-Justine, a tertiary-quaternary care center that mostly serves pediatric patients with SHCN. The experimental group will receive the VR video game Dream designed specifically for this study. It aims at reducing anxiety in children aged 6 to 17 years old by mean of immersive distraction. The VR headset offers children with the ability of viewing the game they are playing in real time while simultaneously obstructing the partial view they would normally have of the procedure. The primary outcome will be assessment of dental fear and anxiety in children using both observation-based proxy assessment with the Venham Anxiety and Behavior Rating Scale (VABRS) and a physiological biomarker such as the level of salivary alpha-amylase. Sociodemographic characteristics, measures of level of satisfaction of parents and healthcare professionals, occurrence of side effects and any deviation from normal procedure length will also be collected. Analysis will be carried out using statistical analysis software SAS (version 9.4; Cary, NC, USA). Descriptive statistics will be conducted for demographic and clinical variables and will be used to present parents and healthcare professionals' satisfaction levels, and also procedural time.

Discussion. The investigators believe that the results of this pilot study will provide a better understanding of the feasibility and effect of VR on DFA in children with SHCN.

DETAILED DESCRIPTION:
Background

Dental fear and anxiety (DFA) is a condition that affects approximately 13.3% to 29.3% of children and adolescents, and is a significant cause of patients avoiding dental care. In children, DFA is also associated with a lower oral-health-related quality of life. Although the etiology of DFA is multifactorial, often stemming from both exogenous and endogenous sources, a previous traumatic dental experience is the most predictive factor for DFA. The majority of DFA experienced by adults stems from poor dental experiences as children. These findings highlight the importance of keeping each dental experience a positive one for pediatric patients. Short term distress during appointments that is not managed properly can accumulate into poor dental experiences, and in turn, reinforcing DFA into adulthood. Long term effects of these poor dental experiences as children can lead patients to avoid seeking proper dental care in the future.

Dental patients with special health care needs (SHCN) are defined as patients requiring additional time and special consideration when receiving treatment due to medical, physical, cognitive or developmental conditions. The population includes children with behaviour (e.g. autism spectrum, anxiety, ADHD), congenital (e.g. trisomy 21, congenital heart disease), developmental (e.g. cerebral palsy), systemic (e.g. childhood cancer, sickle cell disease), or cognitive disorders (eg. intellectual disability). Children with SHCN face more barriers to dental care than the overall population. Barriers include external factors (transportation, cost, inadequate dental facilities) and internal factors (fear and poor tolerance). Many children with SHCN are cared for by dentists in the community, or more often times, in hospital dental clinic settings. They likewise experience more anxiety than those without a disability, which can result in more difficult dental visits. The importance in providing well-rounded care and making each dental visit a positive one for pediatric patients with SHCN is crucial in promoting a good oral health routine, as well as improving their oral health into adulthood.

Understanding and assessing DFA in children is important for delivering successful dental care with high satisfaction in this age group. Among the vast assessment method options available today, self-report assessment, parental proxy assessment, observation-based assessment and physiological assessment are the four major types for children with SHCN. Further, salivary alpha-amylase, an enzyme correlated to both adrenaline and noradrenaline, has also been used as a marker for autonomic nervous system activity and stress.

Factors in the dental setting that trigger DFA include the loud sounds of dental instruments, presence of strangers examining the oral cavity, and the fear of pain. Of these, the anticipation and use of local anesthetic injections are by far the main triggers. Although necessary to provide adequate pain control during certain treatments, local anesthetic injections are uncomfortable. For children, the initial injection combined with the feeling of numbness during the procedure is especially distressing. Pharmacological agents, combined with light to moderate sedation, or general anesthesia can also be considered for non-cooperative patients, but they are often time consuming and at a higher cost as well as generating health risks. Audiovisual distractions such as tablets/TV screens have been used as distraction techniques during dental procedures with overall positive results. However, there is a lack of interactivity of these techniques, and as a result, are not enough to distract children from the stressful procedure. Further, lack of patient cooperation due to DFA often requires dentists treating pediatric populations to end appointments prematurely, and sometimes without completion of the planned procedure. Treating an anxious and fearful patient can also create an environment of stress for the clinician and associated dental team.

Moreover, when treating children with SHCN, extra time and tools are needed to provide comfortable dental care. Depending on the child's diagnosis, many have hypersensitivity to external stimuli such as loud noises, aversion to specific tastes and difficultly straying from usual daily routines. A study by Pagano et al. (2022) showed that the use of augmented reality was well suited for patients with autism spectrum disorder in preparation for their dental visits. Additionally, a systematic review by Cunningham et al. (2021) concluded that virtual reality is a promising tool in dentistry, especially in the population of children with autism spectrum disorder or other special needs.

Aim of the Study

The aims of the study are twofold: (1) assess the feasibility and acceptability of VR immersion as a tool to reduce dental fear and anxiety in pediatric patients with special health care needs undergoing dental procedures and (2) gain insight on parent and healthcare providers' perspectives on the use of VR during dental appointments.

Objectives

The primary research objectives are is to determine:

1. The feasibility and acceptability of VR distraction for children with special needs requiring dental procedures;
2. To compare parent's satisfaction levelshealthcare professionals' satisfaction levels between the VR distraction group and the clinic's standard mounted TV showing cartoons;
3. To observe the preliminary effects of VR distraction in reducing patient anxiety during dental procedures compared to standard non-pharmacological behaviour management.

The secondary objectives of this study are as follows:

1. To compare the occurrence of side effects between the VR distraction group and the clinic's standard mounted TV showing cartoons.
2. To compare dental procedure length between the VR distraction group and the clinic's standard mounted TV showing cartoons
3. To compare the number of retakes of dental procedures due to DFA between the VR distraction group and the clinic's standard mounted TV showing cartoons

MATERIALS AND METHOD

Design

This randomized controlled trial pilot study will follow a parallel design including two groups: a control group (mounted wall TV playing cartoons) and an experimental group (virtual reality intervention during the dental procedure).

Sample and Setting

This pilot will include 20 participants, totalling 10% (10/100) of the expected 200 children to be included in the final study. All participants in this pilot study will be allocated in an equal ratio of 10 per group. Recruitment will be carried out at the dental clinic of the Centre Hospitalier Universitaire Sainte-Justine, a paediatric hospital in Montréal, Canada. This clinic mostly serves patients with special health care needs such as craniofacial abnormalities, autism spectrum disorder, children battling cancer, and others. Pediatric patients with SHCN represents around 80% of the total clientele of this clinic while the rest is comprised of otherwise healthy patients with dental traumas and other dental emergencies. Participants will be identified by the clinic's resident dentist using the scheduling system for upcoming appointments for specific painful dental procedures such as teeth extractions, fillings, and others. The resident dentist will proceed to contact the parents or legal guardian in order to provide information on the study and seek parents' approval ahead of time. An individual independent to the study will review consent with participants and parents. The information and consent form will be signed by one of the parents on the day of the visit.

Randomization and allocation

Randomization will be done through the electronic RedCap system. Allocation to either intervention will be randomized by an independent biostatistician from the URCA (Applied Clinical Research Unit). In order to equalize participants in both arms, permuted block randomization with randomly selected block sizes design will be used to randomize participants to their intervention. Access to the randomization list will only be granted to the biostatistician and allocation will be concealed using RedCap (Research Electronic Data Capture) to reduce selection bias.

Virtual reality and Game Specification

Virtual reality (VR) is defined as an artificial environment which is experienced through sensory stimuli. It is a modern tool that can immerse patients in a "game" or "world." Commonly used in the medical field to help distract patients during unpleasant procedures such as vaccination, cast removal and short bedside interventions, it has proven to be effective at decreasing anxiety and providing a more positive experience for patients. Amongst the limited existing literature, the use of VR to manage anxiety during dental procedures have shown positive results. A recent clinical trial by Alshatrat et al (2022) concluded that VR is an effective tool in reducing anxiety in young children during dental procedures. Moreover, a previous study by Ram et al. (2010) showed that both parent and clinician satisfaction was high using audio-visual glasses as direction for children during dental treatments. However, clinical VR research in pediatric dentistry is limited, especially with special needs populations. VR use in pediatric dentistry offers the potential of an additional non-pharmacologic tool to a clinician's toolbox. A clinical study on the use of VR during dental appointments in pediatric patients with SHCN would allow better understanding on the effect of VR on dental fear and anxiety in this population and facilitate dental procedures.

Designed by Paperplane Therapeutics, Dream is an easy-to-play and immersive VR video game tailored for the paediatric population and approved by a team of health care professionals in paediatric care. The simplified no-success game allows it to be enjoyable no matter the child's video game experience and its point-and-shoot arcade style also allows for easy understanding and fast immersion in the game. Dream was designed specifically for this study with the specific horizontal position in mind needed for dental procedures as well as its eye-tracking navigating system. Dream is designed to be supported by the Pico Neo VR headset.

Children playing the game will be immersed through in a floating gimble that moves from one tropical island to the other. The objective of the game is to throw balls at targets located on the islands such as balloons, trolls, and diamonds in order to gain points. Dream game uses an on-rail feature guiding the child through space with a new eye tracking technology developed within the headset in order to help the child navigate the same way head movement normally would in classic VR, making it easier for dental procedures where head movements are restricted. These features also aim to reduce cybersickness.The preliminary version of the VR headset has been tested in clinic on staff - the size and volume of the headset do not hinder delivery of dental care.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6 to 17 years
* Received the dentist's recommendation to participate
* Required to undergo any dental procedure
* Accompanied by a parent or a legal guardian who can understand, read, and write in either French or English.

Exclusion Criteria:

* Suffer from epilepsy or any other conditions preventing them from using virtual reality (VR).

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
The patient recruitment rates and of completion rate of planned procedures | Patient requirement rates and completion rate of planned procedures will be reported throughout study completion (approx 1 year)
  The feasibility and acceptability of VR distraction for children with special needs requiring dental procedures will be assessed by recording patient recruitment rates and of completion rate of planned procedures.
Parent's or legal guardian's satisfaction | Satisfaction questionnaire is reported by parents immediately following completion of the dental procedure
  Parent's or legal guardian's satisfaction on the intervention and side effects will be assessed using the Visual analog Scale, (0-10, where 0 is very dissatisfied and 10 in very satisfied) and following the recommended question by Pediatric Initiatives on Methods, Measurement and Pain Assessment in Clinical Trials (PedIMMPACT): "Considering anxiety relief, side effects and emotional recovery, how satisfied were you with the intervention used to manage dental fear and anxiety experienced by your child?"
Anxiety | Anxiety scale score is recorded by the operator at the following timepoints: Before the dental procedure to establish baseline; immediately after of completion of dental intervention appointment
  Mean difference in dental fear and anxiety score as measured by proxy using the Venham Anxiety and Behavioral Rating Scale
Healthcare professional's satisfaction | Satisfaction questionnaire is reported by healthcare professional immediately following completion of the dental procedure
  Healthcare professional's satisfaction on the intervention and side effects will be assessed using the Visual Analog Scale, (VAS; ranked from 0-10, where 0 is very dissatisfied and 10 in very satisfied) used to answer the 7-item tailored questionnaire.
Change in Salivary Alpha-Amylase Concentrations before and after dental procedure | Salivary amylase swab will be performed at the following timepoints: Baseline pre-dental procedure; immediately after completion of dental intervention appointment
  Mean difference in salivary alpha-amylase concentration results.

SECONDARY OUTCOMES:
Occurrence of side effects | Any occurence in side effects will be recorded at the following timepoints: baseline pre- dental intervention , during the dental intervention, and immediately after completion of dental intervention appointment
  Recorded as a clinical data. Occurrence of side effects will be collected from arrival on site to discharge from study using a checklist of common side effects experienced while using VR and also related to dental medication.
Length of procedure | The length of the procedure will be noted immediately after completion of the dental intervention appointment
  Recorded as a clinical data. Length of procedure will be measured and collected for every participant and will be compared to average duration for similar procedure that will have been measured prior to the study by the clinic's personnel.
Number of rescheduled of procedures | Any need to reschedule procedures immediately after completion of dental intervention appointment
  Recorded as a clinical data. Rescheduling of procedures in the event where cooperation is impossible.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Le May, PhD, Principal Investigator — St. Justine's Hospital
Locations (1):
- St.Justine's Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cianetti S, Lombardo G, Lupatelli E, Pagano S, Abraha I, Montedori A, Caruso S, Gatto R, De Giorgio S, Salvato R. Dental fear/anxiety among children and adolescents. A systematic review. Eur J Paediatr Dent. 2017 Jun;18(2):121-130. doi: 10.23804/ejpd.2017.18.02.07. PMID 28598183
- [Background] Murad MH, Ingle NA, Assery MK. Evaluating factors associated with fear and anxiety to dental treatment-A systematic review. J Family Med Prim Care. 2020 Sep 30;9(9):4530-4535. doi: 10.4103/jfmpc.jfmpc_607_20. eCollection 2020 Sep. PMID 33209758
- [Background] Luoto A, Lahti S, Nevanpera T, Tolvanen M, Locker D. Oral-health-related quality of life among children with and without dental fear. Int J Paediatr Dent. 2009 Mar;19(2):115-20. doi: 10.1111/j.1365-263X.2008.00943.x. PMID 19250394
- [Background] Beaton L, Freeman R, Humphris G. Why are people afraid of the dentist? Observations and explanations. Med Princ Pract. 2014;23(4):295-301. doi: 10.1159/000357223. Epub 2013 Dec 20. PMID 24356305
- [Background] Humphris G, King K. The prevalence of dental anxiety across previous distressing experiences. J Anxiety Disord. 2011 Mar;25(2):232-6. doi: 10.1016/j.janxdis.2010.09.007. Epub 2010 Sep 19. PMID 20952156
- [Background] Ten Berge M, Veerkamp JS, Hoogstraten J. The etiology of childhood dental fear: the role of dental and conditioning experiences. J Anxiety Disord. 2002;16(3):321-9. doi: 10.1016/s0887-6185(02)00103-2. PMID 12214817
- [Background] Shim YS, Kim AH, Jeon EY, An SY. Dental fear & anxiety and dental pain in children and adolescents; a systemic review. J Dent Anesth Pain Med. 2015 Jun;15(2):53-61. doi: 10.17245/jdapm.2015.15.2.53. Epub 2015 Jun 30. PMID 28879259
- [Background] Oliveira MA, Vale MP, Bendo CB, Paiva SM, Serra-Negra JM. Influence of negative dental experiences in childhood on the development of dental fear in adulthood: a case-control study. J Oral Rehabil. 2017 Jun;44(6):434-441. doi: 10.1111/joor.12513. Epub 2017 May 3. PMID 28386938
- [Background] Koneru A, Sigal MJ. Access to dental care for persons with developmental disabilities in Ontario. J Can Dent Assoc. 2009 Mar;75(2):121. PMID 19267962
- [Background] Yon MJY, Chen KJ, Gao SS, Duangthip D, Lo ECM, Chu CH. An Introduction to Assessing Dental Fear and Anxiety in Children. Healthcare (Basel). 2020 Apr 4;8(2):86. doi: 10.3390/healthcare8020086. PMID 32260395
- [Background] Vacaru RP, Didilescu AC, Sfeatcu R, Tanase M, Munteanu A, Miricescu D, Kaman WE, Brand HS. The Effect of Dental Treatments in Caries Management on Stress and Salivary Protein Levels. J Clin Med. 2022 Jul 27;11(15):4350. doi: 10.3390/jcm11154350. PMID 35893440
- [Background] Morgan AG, Rodd HD, Porritt JM, Baker SR, Creswell C, Newton T, Williams C, Marshman Z. Children's experiences of dental anxiety. Int J Paediatr Dent. 2017 Mar;27(2):87-97. doi: 10.1111/ipd.12238. Epub 2016 Jul 4. PMID 27376925
- [Background] Al-Khotani A, Bello LA, Christidis N. Effects of audiovisual distraction on children's behaviour during dental treatment: a randomized controlled clinical trial. Acta Odontol Scand. 2016 Aug;74(6):494-501. doi: 10.1080/00016357.2016.1206211. Epub 2016 Jul 13. PMID 27409593
- [Background] Alshatrat SM, Sabarini JM, Hammouri HM, Al-Bakri IA, Al-Omari WM. Effect of immersive virtual reality on pain in different dental procedures in children: A pilot study. Int J Paediatr Dent. 2022 Mar;32(2):264-272. doi: 10.1111/ipd.12851. Epub 2021 Jul 5. PMID 34133809
- [Background] Pagano S, Lombardo G, Coniglio M, Donnari S, Canonico V, Antonini C, Lomurno G, Cianetti S. Autism spectrum disorder and paediatric dentistry: A narrative overview of intervention strategy and introduction of an innovative technological intervention method. Eur J Paediatr Dent. 2022 Mar;23(1):54-60. doi: 10.23804/ejpd.2022.23.01.10. PMID 35274543
- [Background] Cunningham A, McPolin O, Fallis R, Coyle C, Best P, McKenna G. A systematic review of the use of virtual reality or dental smartphone applications as interventions for management of paediatric dental anxiety. BMC Oral Health. 2021 May 7;21(1):244. doi: 10.1186/s12903-021-01602-3. PMID 33962624
- [Background] Eijlers R, Utens EMWJ, Staals LM, de Nijs PFA, Berghmans JM, Wijnen RMH, Hillegers MHJ, Dierckx B, Legerstee JS. Systematic Review and Meta-analysis of Virtual Reality in Pediatrics: Effects on Pain and Anxiety. Anesth Analg. 2019 Nov;129(5):1344-1353. doi: 10.1213/ANE.0000000000004165. PMID 31136330
- [Background] McGrath PJ, Walco GA, Turk DC, Dworkin RH, Brown MT, Davidson K, Eccleston C, Finley GA, Goldschneider K, Haverkos L, Hertz SH, Ljungman G, Palermo T, Rappaport BA, Rhodes T, Schechter N, Scott J, Sethna N, Svensson OK, Stinson J, von Baeyer CL, Walker L, Weisman S, White RE, Zajicek A, Zeltzer L; PedIMMPACT. Core outcome domains and measures for pediatric acute and chronic/recurrent pain clinical trials: PedIMMPACT recommendations. J Pain. 2008 Sep;9(9):771-83. doi: 10.1016/j.jpain.2008.04.007. Epub 2008 Jun 17. PMID 18562251
- [Background] Venham LL. The effect of mother's presence of child's response to dental treatment. ASDC J Dent Child. 1979 May-Jun;46(3):219-25. No abstract available. PMID 285948
- [Background] Sahebalam R, Rafieinezhad R, Boskabad M. Comparison of the Efficacy of Jilo Animation Approach versus Conventional Tell-Show-Do (TSD) Technique on Cooperation and Anxiety Levels of Children during Dental Practice: A Randomized Controlled Clinical Trials. J Dent (Shiraz). 2020 Dec;21(4):284-291. doi: 10.30476/dentjods.2020.81897.1001. PMID 33344678
- [Background] Nunna M, Dasaraju RK, Kamatham R, Mallineni SK, Nuvvula S. Comparative evaluation of virtual reality distraction and counter-stimulation on dental anxiety and pain perception in children. J Dent Anesth Pain Med. 2019 Oct;19(5):277-288. doi: 10.17245/jdapm.2019.19.5.277. Epub 2019 Oct 30. PMID 31723668
- [Background] Furlan NF, Gaviao MB, Barbosa TS, Nicolau J, Castelo PM. Salivary cortisol, alpha-amylase and heart rate variation in response to dental treatment in children. J Clin Pediatr Dent. 2012 Fall;37(1):83-7. doi: 10.17796/jcpd.37.1.n32m21n08417v363. PMID 23342572
- [Background] Alaki SM, Safi A, Ouda S, Nadhreen A. Comparing Dental Stress in New Child Patients and Returning Patients Using Salivary Cortisol, Immunoglobulin-A and Alpha- Amylase. J Clin Pediatr Dent. 2017;41(6):462-466. doi: 10.17796/1053-4628-41.6.8. Epub 2017 Sep 22. PMID 28937902
- [Background] AlMaummar M, AlThabit HO, Pani S. The impact of dental treatment and age on salivary cortisol and alpha-amylase levels of patients with varying degrees of dental anxiety. BMC Oral Health. 2019 Sep 6;19(1):211. doi: 10.1186/s12903-019-0901-7. PMID 31492133
- [Background] Chaturvedi Y, Chaturvedy S, Marwah N, Chaturvedi S, Agarwal S, Agarwal N. Salivary Cortisol and Alpha-amylase-Biomarkers of Stress in Children undergoing Extraction: An in vivo Study. Int J Clin Pediatr Dent. 2018 May-Jun;11(3):214-218. doi: 10.5005/jp-journals-10005-1514. Epub 2018 Jun 1. PMID 30131644
- [Derived] Wu W, Le May S, Hung N, Fortin O, Genest C, Francoeur M, Guingo E, St-Arneault K, Sylfra A, Vu AK, Carmel J, Lessard L, Cara-Slavich S, De Koven K, Paquette J, Hoffman H, Asselin ME. Effects of a Virtual Reality Game on Children's Anxiety During Dental Procedures (VR-TOOTH): Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2023 Nov 10;12:e49956. doi: 10.2196/49956. PMID 37948113
- See also: American Academy of Pediatric Dentistry. Management of dental patients with special health care needs. The Reference Manual of Pediatric Dentistry. — https://www.aapd.org/research/oral-health-policies--recommendations/